CLINICAL TRIAL: NCT05434260
Title: The Use of Povidone-iodine Sterile Solution to Reduce Periprosthetic Joint Infections: a Superiority Multicentre Randomized Trial
Brief Title: Surgiphor vs Saline Joints
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Center for Innovation and Research Organization (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Surgiphor01
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Prosthetic-joint Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Surgiphor: sterile povidone iodine irrigation solution (Active Comparator): Surgiphor Wound Irrigation Solution, bottle consisting of sterile 0.5% PVP-I formulation with 0.9% saline, Potassium Iodide, Phosphate Buffer, Vitamin E TPGS
  Interventions: Device: Surgiphor Irrigation Solution
- Sterile saline (Placebo Comparator)
  Interventions: Device: Sterile saline

INTERVENTIONS:
Device: Surgiphor Irrigation Solution — use of Surgiphor wound irrigation solution during surgery
  Arms: Surgiphor: sterile povidone iodine irrigation solution
Device: Sterile saline — Use of sterile saline as a irrigation solution during surgery
  Arms: Sterile saline

SUMMARY:
This study will be an open-label superiority, multicenter, single-blind, controlled randomized clinical trial investing the role of a PVP-I irrigation solution (Surgiphor) in reducing the risk of acute PJI in the 90 days following total hip and knee revision arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥18 years old
2. Male or non-pregnant, non-lactating, postmenopausal or surgically sterilized females
3. Subjects scheduled to undergo total knee or total hip revision for aseptic reasons (per 2018 ICM criteria 5)
4. Subjects provide informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information. Subjects not willing to sign consent form to be randomized must be willing to sign alternate consent form to allow prospective data collection in the non-randomized arm of the study

Exclusion Criteria:

1. Subjects with known allergies to iodine or any other ingredients in Surgiphor
2. Subjects unwilling to sign informed consent
3. Subjects, for health reasons or other, in the opinion of the Investigator, with a life expectancy less than one year, which is the follow-up period of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 868 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of acute prosthetic joint infection | Within 90 days of revision surgery
  Diagnosis of acute prothetic joint infection following aseptic revision surgery

SECONDARY OUTCOMES:
Wound complications | within 1 year of revision surgery
  Diagnosis of wound complication, surgical site infections or other infections within 1 year of surgery

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Arizona, Phoenix, Arizona
  - Lifebridge Health, Baltimore, Maryland
  - University of Missouri, Columbia, Missouri
  - Rothman Institute Orthopaedics, Philadelphia, Pennsylvania